CLINICAL TRIAL: NCT02575365
Title: Effect of Fingolimod on Neurodegeneration, Brain Atrophy and Cognitive Impairment in Relapsing Remitting Multiple Sclerosis Patients
Brief Title: Effect of Fingolimod on Neurodegeneration
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was terminated due to low enrollment.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DTR05
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-10

CONDITIONS: Cognition; Brain Volume Loss
Keywords: RRMS,; Cognition,; brain,; Fingolimod,; Multiple Sclerosis,; neurodegeneration,; Brain atrophy,; gray matter atrophy,; thalamic atrophy,; biomarkers,; BICAMS Battery,
MeSH Terms: conditions — Multiple Sclerosis; Nerve Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fingolimod arm (Experimental): 0.5 mg p.o fingolimod daily
  Interventions: Drug: 0,5 mg Fingolimod

INTERVENTIONS:
Drug: 0,5 mg Fingolimod — 0.5 mg p.o fingolimod daily

SUMMARY:
This was a 24-month, open-label, multicenter study with a single treatment arm design.

Primary objective of this study was:

-To investigate the effects of Fingolimod on cognitive performance in highly active relapsing remitting multiple sclerosis patients

Secondary objectives of this study were:

* To investigate the correlation between the effect of fingolimod on cognitive performances and MRI data.
* To evaluate the effect of fingolimod on biomarkers (24 hydroxy cholesterol, osteopontin and matrix metalloproteinases) related to neurodegeneration
* To investigate the effect of fingolimod on brain gray matter atrophy and thalamic atrophy.

Polulation The hope was to recruit a minimum of 80 relapsing remitting MS (RRMS) patients according to the McDonald criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with RRMS as described in 2010 McDonald criteria (36)
2. Provided written informed consent prior to any intervention
3. Unresponsive to treatment with a beta interferon or glatiramer acetate for a minimum of one year at and at adequate dose and with high disease activity .

   (Unresponsive patients: patients with no changes in relapses, increased relapses, severer relapses with one-year treatment or those who had had at least one relapse during the past one year under previous treatments and one or multiple contrast enhancing lesions in cranial MRI or increased T2 lesions in successive MRIs)
4. EDSS score below 5.5 at screening

Exclusion Criteria:

* 1. Patients with primary or secondary progressive or progressive relapsing MS. 2. Patients with known contraindications for fingolimod treatment. 3. Other coexistent autoimmune diseases including Hashimoto thyroiditis, systemic lupus erythematosus, rheumatoid anthiritis, psoriasis etc.

  4. Patients with any of the following cardiovascular conditions:
  * Resting heart rate < 45 bpm/min
  * Cardiac failure at any time during the first study visit (Class III as per NYHA classification) or significant heart disease as judged by the physician
  * Myocardial infarction during the last 6 months
  * History of Mobitz Type II grade 2 AV block
  * Past or current grade 3 AV block
  * Confirmed history of sick sinus syndrome or sino-atrial heart block
  * arrhythmia requiring current treatment with Class Ia drugs (ajmaline, disopyramid, procainamide, quinidine)
  * hypertension uncontrolled with medication 5. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.

    6. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, detected by urinalysis and confirmed by a positive hCG laboratory test.

    7. Negative for varicella-zoster virus IgG antibodies at screening. Patients who have negative results for varicella-zoster virus IgG antibodies can be included in the study after vaccination for varicella-zoster virus.

    8. Active systemic bacterial, viral or fungal infections, or diagnosis of AIDS, Hepatitis B, Hepatitis C infection defined as a positive HIV antibody, Hepatitis B surface antigen or Hepatitis C antibody tests, respectively 9. History of previous fingolimod therapy 10. Patient who received any of the treatments below:
    1. Corticosteroids or adrenocorticotropic hormone (ACTH) during the last 1 month
    2. Immunosuppressive medications such as azathioprine or methotrexate etc.
    3. Immunoglobulin treatment during the last 3 months
    4. Cladribine, cyclophosphamide, mitoxantrone, natalizumab at any time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Bursa
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Kütahya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned to recruit 80 patients. By the end of the first year, 4 patients have been recruited and the study was stopped due to low enrollment and study results were analyzed.
Period: Overall Study
Arm/Group | Fingolimod Arm
Started | 4
Completed | 0
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Exposed population
Arm/Group | Fingolimod Arm
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race/Ethnicity, Customized [Number; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in The Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) Battery Test at 12 Months
Description: The Brief International Cognitive Assessment for MS ( BICAMS Battery ) includes 3 cognitive tests, 1-Symbol Digit Modalities Test (SDMT, 2-the second edition of the California Verbal Learning Test (CVLT2) and 3-the revised Brief Visuospatial Memory Test (BVMTR).
Time Frame: baseline , month 12.
Population: The trial terminated early because there were only 4 patients who enrolled and only baseline visit was conducted.
Arm/Group | Fingolimod Arm
Number analyzed (Participants) | 0

2. Primary Outcome: Change From Baseline in The Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) Battery Test at 24 Months
Description: The Brief International Cognitive Assessment for MS (BICAMS Battery) includes 3 cognitive tests, 1-Symbol Digit Modalities Test (SDMT, 2-the second edition of the California Verbal Learning Test (CVLT2) and 3-the revised Brief Visuospatial Memory Test (BVMTR).
Time Frame: baseline and month 24
Population: The trial terminated early because there were only 4 patients who enrolled and only baseline visit was conducted.
Arm/Group | Fingolimod Arm
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in PASAT Test
Description: The Paced Auditory Serial Addition Test (PASAT) has been widely used in MS trials and it is considered to be a measure of sustained attention, divided attention, concentration, and information processing speed.
Time Frame: baseline ,months 6, month 12 and month 24
Population: The trial terminated early because there were only 4 patients who enrolled and only baseline visit was conducted.
Arm/Group | Fingolimod Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Stroop Test
Description: The Stroop Color and Word Test assesses cognitive processing and provides valuable diagnostic information on brain dysfunction, cognition, and psychopathology
Time Frame: baseline, month 6, month 12 and month 24
Population: The trial terminated early because there were only 4 patients who enrolled and only baseline visit was conducted.
Arm/Group | Fingolimod Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Brain Gray Matter Atrophy and Thalamic Atrophy
Description: MRI scans will be obtained by using 1,5T MRI for measuring gray matter atrophy and thalamic atrophy and a standard scanning protocol will be used for MRI in all centers.
Time Frame: baseline, month 6, month 12, month 18 and month 24
Population: The trial terminated early because there were only 4 patients who enrolled and only baseline visit was conducted.
Arm/Group | Fingolimod Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Serum Levels of 24S-hydroxycholesterol (24OHC) , Osteopontin and Matrix Metalloproteinases (and Also MMPI's)
Description: Serum samples will be collected at baseline and at months 6, 12 and 24 from each participant after evaluation for inclusion and exclusion criteria for measurement of 24 hydroxy cholesterol, osteopontin and matrix metalloproteinases (including MMPI's).
Time Frame: baseline, month 6, month , month 12 and month 24
Population: The trial terminated early because there were only 4 patients who enrolled and only baseline visit was conducted.
Arm/Group | Fingolimod Arm
Number analyzed (Participants) | 0

7. Secondary Outcome: the Correlation Between Effect of Fingolimod on Cognitive Performances and Brain Atrophy (Gray Matter Atrophy and Thalamic Atrophy) by Comparing Baseline and Month 24.
Description: Correlation between effect of fingolimod on cognitive performances based on cognitive tests and brain atrophy based on MRI assessments will be explored.
Time Frame: baseline, month 24
Population: The trial terminated early because there were only 4 patients who enrolled and only baseline visit was conducted.
Arm/Group | Fingolimod Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit, up to approximately 11 months.
Arm/Group | Fingolimod Arm
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fingolimod Arm (N=4)
Headache (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was terminated due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT02575365/Prot_SAP_000.pdf